CLINICAL TRIAL: NCT03719209
Title: Using Virtual Reality to Foster Engagement, Understanding, and Knowledge in Patients With Gastrointestinal Disease and Their Families
Brief Title: Using Virtual Reality for Patients With Gastrointestinal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Klick Health (Unknown)
Responsible Party: Principal Investigator, Michael Docktor, Attending Physician, Division of Gastroenterology, Hepatology, and Nutrition, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P00024632
Record Dates: First submitted 2018-10-07; First posted 2018-10-25 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2018-10

CONDITIONS: Gastrointestinal Disease; Inflammatory Bowel Diseases
Keywords: Crohns disease; Patient Education; Ulcerative Colitis; Celiac; Ulcer; Polyp; Gastrointestinal bleeding; Inflammatory Bowel Disease; Virtual Reality
MeSH Terms: conditions — Gastrointestinal Diseases; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Celiac Disease; Ulcer; Polyps; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Practice (Placebo Comparator): Patients and families will be shown images of their endoscopic procedure per standard practice.
  Interventions: Other: Standard Practice
- Virtual Reality (Experimental): Patients and families will be showed the results of their endoscopic procedure via a virtual reality application called HealthVoyager, in addition to standard practice images.
  Interventions: Other: HealthVoyager

INTERVENTIONS:
Other: HealthVoyager — HealthVoyager is a virtual reality application that allows providers to create customized representations for patients and share the results of endoscopic procedures via an interactive platform. The app can show both normal and abnormal endoscopic findings and anatomy. Families will also receive a web link so that they may access the procedure results via the app at home on their smartphone or tablet.
  Arms: Virtual Reality
Other: Standard Practice — Patients and families will receive handouts with printed images of their endoscopic findings, as per standard practice at Boston Children's Hospital.
  Arms: Standard Practice

SUMMARY:
The primary aim of this study is to evaluate the effect and impact of a technology which creates a virtual reality (VR), personalized representation of a patient's endoscopic findings in comparison our standard practice (SP). Our study will compare the level of knowledge, understanding and satisfaction the patient and family have between those receiving SP and those receiving both SP and VR.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8-25 years of age who are willing and able to participate
* Patients who recently had an endoscopic procedure at Boston Children's Hospital

Exclusion Criteria:

* Patients who are unable to provide consent due to age or developmental status

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Patient and family knowledge, understanding, and satisfaction | 1 month
  Our study will measure the levels of patient and family engagement using a survey designed specifically for the study. The survey is at a roughly 3rd grade reading level and includes approximately 10 questions with answers on a Likert scale. The internally designed survey will specifically measure patient and family opinions on learning about the results of their procedure, as well as objective anatomical knowledge. The minimum score for each question is a 1, designating "Strongly disagree." The maximum score for each question is a 10, designating "Strongly agree." Thus, higher scores represent better outcomes.

SECONDARY OUTCOMES:
Longitudinal Medication Adherence | up to 5 years
  Medication Adherence will be assessed via retrospective chart review and medication refill data.
Longitudinal Readmission Rate | up to 5 years
  Readmission rates will be measured via retrospective chart review and hospital admission data.
Patient Satisfaction Scale | 1 month
  The Patient Satisfaction Scale (Hojat et al., 2011) will be used to measure patient satisfaction. The Patient Satisfaction Scale is a validated survey with 10 questions. Respondents can answer 1 through 7 for each question. 1 represents "Strongly Disagree" while 7 represents "Strongly Agree." Higher score represent better outcomes in this scale.
Client Satisfaction Questionnaire | 1 month
  The Client Satisfaction Questionnaire (Larsen et al., 1979) will measure client satisfaction. The questionnaire has 8 questions with 4 possible answers for each question. A 4 represents the best possible outcome; a 1 represents the worst possible outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palanica A, Leier M, Lee A, Fossat Y, Docktor MJ. Enhancing the Patient Experience for Individuals Undergoing Endoscopic Procedures Using Virtual Reality. J Pediatr Gastroenterol Nutr. 2020 Mar;70(3):341-343. doi: 10.1097/MPG.0000000000002577. PMID 31789778